CLINICAL TRIAL: NCT00860834
Title: Parents, Pediatricians, and Telephone Coaches Partner to Improve Control of Asthma
Brief Title: Telephone Coaches to Improve Control of Asthma in Children ( PARTNER) Study)
Acronym: PARTNER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jane Garbutt, MD, Associate Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 634; R01HL072919 (NIH); R01HL072919-06 (NIH)
Record Dates: First submitted 2009-03-10; First posted 2009-03-12 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Asthma
Keywords: Consumer Participation; Telephone Coaching Program
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Pediatricians and parents of children with asthma will participate in the asthma coaching program.
  Interventions: Behavioral: Asthma Coaching Program
- 2 (Active Comparator): Children of parents enrolled in the study will receive usual asthma care from their pediatrician.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Asthma Coaching Program — Parents will have access to an asthma coach for 12 months. Telephone calls between parents and coaches will occur anywhere from once a week to once a month.
  Arms: 1
Behavioral: Usual Care — Children of parents enrolled in the study will receive the normal asthma care that their pediatricians usually provide.
  Arms: 2

SUMMARY:
Parents of children with asthma must work with their child's pediatrician to ensure that their child's asthma is managed well. Asthma coaches are one way to facilitate and support the relationship between parents and pediatricians. This study will evaluate whether access to a 12-month telephone asthma coaching program for parents is an effective way to improve asthma outcomes in children.

DETAILED DESCRIPTION:
Asthma is the most common long-term disease among children. Each year, most children with asthma will have at least one asthma exacerbation, experience asthma symptoms on approximately 100 days, and miss 4 days of school because of asthma. Surveys of primary care physicians (PCPs) and asthma patients have indicated that asthma care is episodic, effective asthma controller medications are underused, and few PCPs provide self-management education or support for parents of children with asthma. Previous research showed that when an asthma coach worked with parents of children from low-income, urban neighborhoods, there were multiple benefits: improved self-management behaviors, reduced asthma hospitalizations, and improved rates of follow-up with a PCP after an emergency department visit for asthma symptoms. In this study, researchers will evaluate the effectiveness of an asthma coach program in a larger, general asthma population. Trained asthma coaches will work with parents of children with asthma to provide education about the goals of asthma care, and they will encourage and facilitate an active partnership between the family and PCP to enhance asthma care and improve self-management behaviors. Study researchers will then evaluate the effectiveness of this program at improving asthma control and quality of life among children with asthma. The cost effectiveness of the program will also be analyzed.

This study will enroll pediatricians and parents of children between 5 and 12 years old who have persistent asthma. Pediatricians will be randomly assigned to either the asthma coach program or usual care. All pediatricians will receive access to the Education in Quality Improvement for Pediatric Practice (eQIPP) module for asthma care provided by the American Academy of Pediatrics. They will also receive articles about effective doctor-parent communication on asthma and asthma billing practices. In addition, pediatricians taking part in the asthma coach program will attend two meetings to learn about asthma coaching and how the program can be implemented into their practice. For 12 months, an asthma coach will work directly with the parents of children who see doctors participating in the asthma coaching group. Telephone calls with the asthma coach will be arranged at times convenient for the parent and will occur anywhere between once a week to once a month. At Months 12 and 24, about 40 parents of children in each pediatrician's practice will participate in telephone interviews and their children's medical charts will be reviewed to assess asthma control, asthma-related quality of life factors, and urgent care events.

ELIGIBILITY:
Inclusion Criteria for Pediatricians:

* Affiliated with St. Louis Children's Hospital and/or Washington University in St. Louis
* Provides asthma care for at least 40 asthmatic children from the target population

Inclusion Criteria for Parents:

* Has a child who is between 3 and 12 years old with persistent asthma and who is cared for by a study pediatrician

Exclusion Criteria for Pediatricians:

* Spends less than 50% of their time in general pediatrics
* Is an asthma specialist (allergist or pulmonary specialist)
* Another physician in their practice is participating in the study

Exclusion Criteria for Parents:

* Their asthmatic child is less than 3 years old or is 13 years or older at the time of study entry
* Their child has not had a physician diagnosis of asthma before study entry
* Their child has a significant comorbid condition
* Cannot speak English
* Does not have a phone

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 984 (Actual)
Dates: Start 2008-08 (Actual); Primary Completion 2013-05-03 (Actual); Study Completion 2014-05-03 (Actual)

PRIMARY OUTCOMES:
Asthma control | Measured at Months 12 and 24
Asthma-related quality of life | Measured at Months 12 and 24
Urgent care events | Measured at Months 12 and 24

SECONDARY OUTCOMES:
Adherence to guideline-recommended asthma maintenance care behaviors | Measured at Months 12 and 24
Cost effectiveness | Measured at Months 12 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Jane M. Garbutt, MB, ChB, Principal Investigator — Washington University School of Medicine; Robert Strunk, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Garbutt JM, Highstein G, Yan Y, Strunk RC. Partner randomized controlled trial: study protocol and coaching intervention. BMC Pediatr. 2012 Apr 2;12:42. doi: 10.1186/1471-2431-12-42. PMID 22469168
- [Derived] Garbutt JM, Yan Y, Highstein G, Strunk RC. A cluster-randomized trial shows telephone peer coaching for parents reduces children's asthma morbidity. J Allergy Clin Immunol. 2015 May;135(5):1163-70.e1-2. doi: 10.1016/j.jaci.2014.09.033. Epub 2014 Oct 30. PMID 25445827